CLINICAL TRIAL: NCT02882750
Title: Curative Treatment Modalities of Early Stages Non-Small Cell Lung Cancer: Effect on Patient Reported Outcomes of Video Assisted Thoracoscopic (VATS) Resection and Stereotactic Ablative Body Radiotherapy (SABR)
Brief Title: Effect on Patient Reported Outcomes of VATS and SABR (LILAC)
Acronym: LILAC
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: Yorkshire Cancer Research (Other); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Galina Velikova, Prof of Clinical Oncology, University of Leeds
Other Study IDs: L399
Record Dates: First submitted 2016-07-07; First posted 2016-08-30 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Lung Cancer
Keywords: Lung Cancer; Quality of Life; VATS; SABR
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Surgical Patients: Early stage NSCLC patients submitted to Surgical Resection
  Interventions: Other: EORTC QLQ-C30 (version 3.0).; Other: PS Q18; Other: Decision Self-Efficacy Scale
- SABR Patients: Early stage NSCLC patients submitted to SABR
  Interventions: Other: EORTC QLQ-C30 (version 3.0).; Other: PS Q18; Other: Decision Self-Efficacy Scale

INTERVENTIONS:
Other: EORTC QLQ-C30 (version 3.0). — Quality of Life Questionnaire
Other: PS Q18 — Patients Satisfaction Questionnaire
Other: Decision Self-Efficacy Scale — Questionnaire

SUMMARY:
This study will monitor the effect on patients reported outcomes (PROMs) of VATS resection and SABR for NSCLC delivered at the Leeds Cancer Centre The investigator will support with this information the Shared Decision Making (SDM) process.

300 consecutive patients will be followed up from prior the treatment to 12 months afterwards, administering multiple questionnaires (EORTC QLQ C-30 and LC-13, PSQ-18, Decision Self-Efficacy Scale) by a remote web-based system.

Deliverable:

1. Differences after VATS resections or SABR in terms of physical and psychological symptoms, quality of life and satisfaction
2. Patient perspectives of the Shared Decision Making Process.

DETAILED DESCRIPTION:
1. Methods

   Aim and Objectives

   This study aims to describe the trajectory of lung cancer patients HRQoL, symptoms and functions following VATS or SABR treatment for Stage I-II NSCLC and to determine the feasibility and patient acceptability of online self-reporting of PROMs.

   Specific objectives of the study include:
   * To compare changes before and after treatment of patient reported outcomes (HRQOL and Patient Satisfaction) after VATS lung resections or SABR in early stage lung cancer patients.
   * To correlate clinical outcomes (complications and AEs) with Quality of Life in order to find objective predictors of major decline in patient reported outcomes.
   * To identify specific factors, which have influenced the personal choice between the treatments (Decision Self-Efficacy Scale)
   * Establish recruitment and attrition rates and adherence to PROMs reporting during the study
   * To describe patient choice of electronic vs paper questionnaires
   * To explore implementation issues through patient and staff interview.
2. Design

This is an observational prospective longitudinal study with repeated measures (PROMs), employing a convenience sample of consecutive patients planned to have VATS resections or SABR for stages I-II of NSCLC. Outcomes measures will be collected prior to treatment and 1,3,6,12 months afterwards, administering the questionnaires by the remote web-based system. Paper administration will be offered to patients without Internet access.

Sample size considerations

Last year 100 pre-surgical quality of life questionnaires have been collected in 5 months from outpatients' clinic at Leeds Cancer Centre (LCC). For longitudinal studies involving regular PROMs, the investigators typically see 70% consent rate and 30-35% attrition over 3 months24. Therefore the investigators expectations are to be able to recruit 200 VATS and 50 SABR patients recruiting over 12 months with 12 months of follow-up.

In order to detect a minimum difference of 10% from the baseline value and standard deviation of the EORTC QLQ-C30 Global Health Scale scale (as measured in our historical cohort of 115 anatomic lung resections), with a alfa level of 0.05 and statistical power of 90%, a sample size of 115 patients in the surgical arm was estimated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and over.
* Diagnosis of NSCLC either from histology or MDT/Tumour Board agreement on >95% likelihood of diagnosis based on radiological evidence or both.
* Decision for either surgery or SABR
* Able to give informed consent.
* Able to understand the language of the questionnaire.
* There will be no limit on performance status.

Exclusion Criteria:

* Advanced diseases (III-IV stages).
* Patient included in other HRQoL study, which may increase patient burden and bias the answer of the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage Non-Small Cell Lung Cancer patients
Sampling Method: Probability Sample
Enrollment: 244 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-04-09 (Actual); Study Completion 2019-06-06 (Actual)

PRIMARY OUTCOMES:
Patients Reported Outcomes | 12 months
  Quality of life (EORTC QLQ-C30 and LC13 questionnaire)

SECONDARY OUTCOMES:
Decision self-efficacy scale | 3 months
  Patient perspectives of the Shared Decision Making Process.
Patient Acceptability | 12 months
  Patient acceptability explored through interviews
Clinician Acceptability | 12 months
  clinician acceptability explored through interviews
Patients satisfaction | 1 month
  patients satisfaction of the care received (PSQ-18 Patient satisfaction questionnaire)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pompili C, Franks KN, Brunelli A, Hussain YS, Holch P, Callister ME, Robson JM, Papagiannopoulos K, Velikova G. Patient reported outcomes following video assisted thoracoscopic (VATS) resection or stereotactic ablative body radiotherapy (SABR) for treatment of non-small cell lung cancer: protocol for an observational pilot study (LiLAC). J Thorac Dis. 2017 Aug;9(8):2703-2713. doi: 10.21037/jtd.2017.07.35. PMID 28932579